CLINICAL TRIAL: NCT02376647
Title: ART-3 Pilot: A Randomized Controlled Trial to Assess the Feasiblity of a Driving Pressure Limited Ventilation vs.Standard Strategy in Patients Without ARDS
Brief Title: ART-3 Pilot - Driving Pressure Limited Ventilation for Patients Without ARDS (ART3pilot)
Acronym: ART-3pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained so far. Project was halted.
Sponsor: Hospital do Coracao (Other)
Collaborators: Brazilian Research in Intensive Care Network (BRICNet) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-3pilot; ART-3pilot (Other Grant/Funding Number: Hospital do Coração)
Record Dates: First submitted 2015-02-13; First posted 2015-03-03 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Mechanical Ventilation; Acute Respiratory Distress Syndrome
Keywords: Patients; ARDS diagnosis
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving pressure limited ventilation (Experimental): Driving pressure limited ventilation (≤13cmH2O)
  Interventions: Other: Driving pressure limited ventilation
- Conventional ventilation (Active Comparator): Mechanical ventilation with limited tidal volume (8mL/kg of predicted body weight) and plateau pressure (≤30cmH2O)
  Interventions: Other: Conventional ventilation

INTERVENTIONS:
Other: Driving pressure limited ventilation — Investigators will use volume controlled (or pressure support ventilation) and adjust tidal volume between 3 and 8 mL/Kg of predicted body weight in order to achieve a driving pressure of 13 cmH2O. The respiratory rate will be titrated to achieve a pH between 7.30 and 7.45 (maximum respiratory rate is 50 breathings per minute). Investigators will not limit plateau pressure in this arm.
  Once a daily the investigators will assess the target tidal volume that generates a driving pressure of 13cmH2O. The patient should be sedated and without spontaneous efforts during this assessment.
  Arms: Driving pressure limited ventilation
Other: Conventional ventilation — Investigators will use volume controlled or pressure support ventilation, tidal volume ≤8 mL/kg of predicted body weight and plateau pressure limited to 30 cmH2O.The respiratory rate will be titrated to achieve a pH between 7.30 and 7.45 (maximum respiratory rate is 35 breathings per minute).
  Arms: Conventional ventilation

SUMMARY:
This is a multicenter randomized controlled pilot trial to investigate the feasibility of a driving pressure limited mechanical ventilation strategy compared to a conventional strategy in patients without acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Mechanical ventilation has the potential to produce or worsen alveolar injury. Driving pressure is the difference between plateau pressure and PEEP. Evidence from observational studies suggests that elevated driving pressure is the main independent determinant of ventilator-induced lung injury, however clinical trials are needed to establish whether targeting low driving pressures can improve clinical outcomes in patients without acute respiratory distress syndrome (ARDS).

Thus, ART-3 pilot is a multicenter randomized controlled trial to assess the feasibility of a driving pressure limited mechanical ventilation strategy compared to a conventional strategy in patients without ARDS. Patients considered to this trial are those in mechanical ventilation for less than 72 hours without diagnosis of ARDS. We will exclude patients with less than 18 years old; contraindication to hypercapnia such as intracranial hypertension or recent acute coronary syndrome; patients in which a high probability of death within 24 hours is anticipated and patients under exclusive palliative care. Eligible patients will be randomized to the driving pressure limited ventilation strategy or conventional strategy (tidal volume of 8 mL/kg of predicted body weight). The primary outcome is driving pressure between days 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients on invasive mechanical ventilation for less than 72 hours and without diagnosis of ARDS, and no perspective of extubation in 24 hours.

Exclusion Criteria:

* Less than 18 years old
* Presence of any contraindication to hypercapnia as suspected or confirmed intracranial hypertension or recent (<7 days) acute coronary syndrome.
* Patients in which a high probability of death within 24 hours is anticipated.
* Patients under exclusive palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Mean driving pressure between Day 1 and Day 3 | From Day 1 to Day 3 after randomization

SECONDARY OUTCOMES:
Rate of investigators adering to study procedures | Days 1 to 7
Rate of driving pressure equal or lower than 13 cmH2O | Days 1 to 3 after randomization
Mean of positive end expiratory pressure (PEEP) from day 1 to 7 | Days 1 to 7
Mean tidal volume from day 1 to 7 | Days 1 to 7
Mean static compliance of the respiratory system from day 1 to 7 | Days 1 to 7
Mean plateau pressure from day 1 to 7 | Days 1 to 7
Mean driving pressure from day 1 to 7 | Days 1 to 7
Mean respiratory rate from day 1 to 7 | Days 1 to 7
Number of patients with barotrauma | Days 1 to 7
Mean of severe acidosis (pH <7.1) | Days 1 to 7
Number of patients with other adverse events | Days 1 to 7
Lenght of stay in intensive care unit | Patients will be followed during the period of ICU stay, an expected average of 28 days
Lenght of stay in hospital | Patients will be followed during the period of hospital stay, an expected average of 28 days
Number of mechanical ventilation free days from day 0 to day 28 | From day 0 to day 28
ICU mortality | Patients will be followed during the period of hospital stay, an expected average of 28 days
In-hospital mortality | Patients will be followed during the period of hospital stay, an expected average of 28 days
28-day survival | From day 0 to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, PhD, Study Chair — Hospital do Coração(Heart Hospital)
Locations (1):
- Alexandre Biasi Cavalcanti, São Paulo, São Paulo, Brazil